CLINICAL TRIAL: NCT04388189
Title: Leveraging EEG for Antidepressant Prediction With Duloxetine and Bupropion (LEAP-DB): A Multicenter, Randomized, Blinded Outcome Study of EEG-guided Treatment With Duloxetine Versus Bupropion in Adults With Major Depressive Disorder
Brief Title: Leveraging EEG for Antidepressant Prediction With Duloxetine and Bupropion
Acronym: LEAP-DB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAP-DB
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; EEG; Biomarker; Antidepressant; Duloxetine; Bupropion
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine (Experimental): Duloxetine 60 mg daily for 8 weeks
  Interventions: Drug: Duloxetine
- Bupropion (Active Comparator): Bupropion 150-450 mg daily for 8 weeks
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Duloxetine — FDA approved antidepressant
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Bupropion — FDA approved antidepressant
  Other Names: Wellbutrin
  Arms: Bupropion

SUMMARY:
The LEAP-DB study will be conducted to validate the utility of EEG biomarkers as an aid to antidepressant treatment selection in adults with MDD.

DETAILED DESCRIPTION:
The LEAP-DB study is an 8-week, multicenter, randomized, blinded study to evaluate the performance of EEG-based biomarkers in predicting treatment outcome. Study participants will be randomized in a 1:1 ratio to receive either duloxetine or bupropion and followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 22 or older at the time of informed consent.
* Diagnosis of Major Depressive Disorder (MDD) based on the Structured Clinical Interview for DSM-5 for depression.
* Moderate or severe depression on DSM-5 depression criteria items, as assessed by a score of 10 or more on the Patient Health Questionnaire (PHQ-9)
* Has not taken either study medications (duloxetine, bupropion) in the current episode
* Has not received electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or esketamine treatment in the current episode
* Provision of personally signed and dated written informed consent prior to any study procedures
* Agrees to, and is eligible for all biomarker assessments (EEG, neurocognitive testing, activity and sleep monitoring, genetic testing)
* Fluent in English
* Ability to complete all assessments independently
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Diagnosis of bipolar disorder or a psychotic disorder based on the Structured Clinical Interview for DSM-5.
* Concurrent use of antipsychotics or mood stabilizers
* Use of hypnotics, anxiolytics or opiate pain medications greater than three days per week and unable to reduce use to three or fewer days per week on an as needed basis
* Pregnant or breastfeeding
* Severe impediment to vision, hearing, comprehension, and/or hand movement that interferes with study tasks
* Active substance use that interferes with ability to consent and/or complete assessments
* Any contraindication to EEG (e.g. requiring high concentration oxygen)
* Employees/family of employees of clinic site
* Participation in another research study that began within less than 2 months prior to the first study visit

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Response rate on the 16-item patient-reported Quick Inventory of Depressive Symptoms (QIDS-SR) at the week 8 endpoint as a function of biomarker score | 8 weeks
  The Quick Inventory of Depressive Symptomatology (QIDS-SR) is a 16 item self-report scale that measures depressive symptoms. The QIDS assesses the severity of all DSM-V criterion items required to diagnose a major depressive episode. It asks the patient to rate each of 16 items on a scale from 0 to 3. Additionally, it states the frequency and severity of symptoms that patients should consider while responding to items in the survey. Each item in the survey asks about depressive symptoms that the patient may have experienced in the past seven days.

SECONDARY OUTCOMES:
Percentage decrease in depressive symptoms on the QIDS-SR at the week 8 endpoint as a function of biomarker score | 8 weeks
  Quick Inventory of Depressive Symptoms (QIDS-SR)
Absolute score decrease from baseline to the week 8 endpoint on the QIDS-SR as a function of biomarker score | 8 weeks
  Quick Inventory of Depressive Symptoms (QIDS-SR)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Keller, MD, PhD, Study Director — Alto Neuroscience

IPD SHARING:
Plan to Share IPD: Undecided